CLINICAL TRIAL: NCT04079296
Title: A Phase 1/2 Open-label Study Investigating the Safety, Tolerability and Efficacy of ASP7517 in Subjects With Relapsed/Refractory Acute Myeloid Leukemia (AML) and Relapsed/Refractory Higher Risk Myelodysplastic Syndrome (MDS)
Brief Title: A Study Investigating the Safety, Tolerability and Efficacy of ASP7517 in Subjects With Relapsed/Refractory Acute Myeloid Leukemia (AML) and Relapsed/Refractory Higher Risk Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 7517-CL-0101
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome
Keywords: ASP7517; Safety; Efficacy; Tolerability
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Escalation (Phase 1): ASP7517 1x10^6 cells/mL (Experimental): Participants with Relapsed/Refractory Acute Myeloid Leukemia (R/R AML) and R/R higher risk Myelodysplastic Syndrome (MDS) received intravenous (IV) infusion of ASP7517 (human embryonic kidney cell [HEK293] transfected with encoding target WT-1) at a dose of 1x10^6 cells/milliliters (mL) at 4 to 6 mL/minute infusion rate on day 1 of each cycle for 2 doses (1 cycle= 28 days).
  Interventions: Biological: ASP7517
- Dose Escalation (Phase 1): ASP7517 1x10^7 cells/mL (Experimental): Participants with R/R AML and R/R higher risk MDS received IV infusion of ASP7517 (HEK293 transfected with encoding target WT-1) at a dose of 1x10^7 cells/mL at 4 to 6 mL/minute infusion rate on day 1 of each cycle for 2 doses (1 cycle= 28 days).
  Interventions: Biological: ASP7517
- Dose Escalation (Phase 1): ASP7517 1x10^8 cells/mL (Experimental): Participants with R/R AML and R/R higher risk MDS received IV infusion of ASP7517 (HEK293 transfected with encoding target WT-1) at a dose of 1x10^8 cells/mL at 4 to 6 mL/minute infusion rate on day 1 of each cycle for 2 doses (1 cycle= 28 days).
  Interventions: Biological: ASP7517
- Dose Expansion (Phase 2: AML): ASP7517 1x10^8 cells/mL (Experimental): Participants with R/R AML received IV infusion of ASP7517 (HEK293 transfected with encoding target WT-1) at a dose of 1x10^8 cells/mL at 4 to 6 mL/minute infusion rate on day 1 of each cycle for 6 doses (1 cycle= 28 days).
  Interventions: Biological: ASP7517
- Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 cells/mL (Experimental): Participants with R/R higher risk MDS received IV infusion of ASP7517 (HEK293 transfected with encoding target WT-1) at a dose of 1x10^8 cells/mL at 4 to 6 mL/minute infusion rate on day 1 of each cycle for 6 doses (1 cycle= 28 days).
  Interventions: Biological: ASP7517

INTERVENTIONS:
Biological: ASP7517 — Intravenous (IV)

SUMMARY:
The purpose of this study was to evaluate the safety and tolerability and to determine the recommended phase 2 dose (RP2D) and/or the maximum tolerated dose (MTD) of ASP7517.

This study also evaluated the clinical response of ASP7517 as well as other measures of anticancer activity of ASP7517.

DETAILED DESCRIPTION:
This study consisted of 2 parts: phase 1 dose escalation and phase 2 dose expansion.

Phase 1 Dose Escalation:

Approximately 18 subjects with either relapsed/refractory (R/R) AML or R/R higher risk MDS were enrolled. Participants received 2 single doses of ASP7517 via intravenous infusion. Dosing occured on day 1 of each cycle. Each cycle was defined as 28 days with a total of 2 treatment cycles.

Participants were managed under hospitalization for at least 7 days during the first cycle of the dose escalation phase. In addition, prior to hospital discharge, participant safety was ensured by performing medical tests and procedures listed on day 7 of cycle 1 and tests considered clinically necessary to evaluate the participant's general condition and adverse event (AE) resolution. The participant was also followed on an outpatient basis on planned visits during cycles 1 and 2 after hospital discharge during the dose limiting toxicity (DLT) assessment period to closely monitor any AEs. Participants were hospitalized days 1 to 7 during cycle 2.

Phase 2 Dose Expansion:

Approximately 104 participants per dose level were enrolled. Each dose level enrolled up to 52 R/R AML participants and up to 52 R/R higher risk MDS participants. Both groups of participants were enrolled in parallel and independently. The number of dose levels investigated during phase 2 were based upon the data from phase 1. When escalation and expansion cohorts were both open for enrollment, enrollment into escalation cohorts took priority such that participants who were eligible for both were preferentially enrolled in the escalation cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Subject diagnosed with R/R AML or R/R higher risk MDS is defined as:

  * R/R AML: Morphologically documented primary or secondary AML by the WHO criteria (2016); and refractory to at least 2 cycles of induction chemotherapy/not a candidate for re-induction or relapsed after achieving remission with a prior therapy; and received all standard therapies including targeted therapies (unless the therapy is contraindicated or intolerable) which are known to provide clinical benefit in the opinion of the treating investigator; and received salvage therapy or is not a candidate for salvage therapy.
  * R/R higher risk MDS: Has MDS by the WHO criteria (2016); and either relapsed after achieving remission or refractory to standard therapies, including ≥ 4 cycles of hypomethylating agents (unless the therapy is contraindicated or intolerable); and is classified as higher risk MDS with a score of > 3.5 by Revised International Prognostic Scoring System (IPSS-R) in MDS.
* Subject has an Eastern Cooperative Oncology Group performance status of ≤ 2.
* Subject must meet the following criteria as indicated on the clinical laboratory tests during screening period:

  * Serum aspartate aminotransferase and alanine aminotransferase ≤ 2.5 × upper limit of normal (ULN).
  * Serum total bilirubin ≤ 1.5 × ULN.
  * Serum creatinine ≤ 1.5 × ULN or an estimated glomerular filtration rate of > 50 mL/min as calculated by the Modification of Diet in Renal Disease equation.
  * Platelets ≥ 50,000/μL at cycle 1 day 1 (C1D1) in the dose escalation cohorts only.
* Subject has a life expectancy of ≥ 12 weeks at the time of screening.
* Subjects with AML must have peripheral blood absolute blast count of < 20,000/μL at C1D1. Note: Blast count can be controlled by hydroxyurea during screening period.
* Female subject is not pregnant and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP).
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 180 days after final study treatment administration.
* Female subject must agree not to breastfeed starting at screening and throughout the study period and for 180 days after the final study treatment administration.
* Female subject must not donate ova starting at first dose of investigational product (IP) and throughout the study period and for 180 days after final study treatment administration.
* Male subject with female partner(s) of childbearing potential (including breastfeeding partner) must agree to use contraception throughout the treatment period and for 180 day after final study treatment administration.
* Male subject must not donate sperm during the treatment period and for 180 days after the final study treatment administration.
* Male subject with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 180 days after final study treatment administration.
* Subject agrees not to participate in another interventional study while receiving study treatment in the present study.

Exclusion Criteria:

* Subject was diagnosed with acute promyelocytic leukemia.
* Subject has breakpoint cluster region-Abelson-positive leukemia (BCR-ABL).
* Subject has persistent non-hematological toxicities of ≥ grade 2 (National Cancer Institute's Common Terminology Criteria for Adverse Events [NCI-CTCAE], version 5.0), with symptoms and objective findings from prior AML or MDS treatment (including chemotherapy, kinase inhibitors, immunotherapy, experimental agents, radiation or surgery).
* Subject has received any of the following therapies:

  * Systemic immunomodulators or immunosuppressive drugs including steroids ≤ 28 days prior to C1D1 (steroids can be used if not intended for treatment of AML or MDS; steroids for AML/MDS related symptoms can be used at low doses [less than 10 mg/day dexamethasone]).
  * Cytotoxic agents (except hydroxyurea given for controlling blast cells) ≤ 28 days prior to C1D1.
  * Investigational products for the treatment of AML or MDS within 5 half-lives prior to screening visit.
  * Hematopoietic stem cell transplant (HSCT).
  * Radiation therapy ≤ 28 days prior to C1D1.
* Subject has clinically active nervous system leukemia.
* Subject has active or prior documented autoimmune or inflammatory disorders requiring systemic treatment.
* Subject has ongoing, untreated malignancy with the exception of the following:

  * Subjects with treated non-melanoma skin cancer, in situ carcinoma or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed.
  * Subjects with organ-confined prostate cancer with no evidence of recurrent or progressive disease are eligible if hormonal therapy has been initiated or the malignancy has been surgically removed or treated with definitive radiotherapy.
* Subject with left ventricular ejection fraction of < 45% on echocardiogram or multigated acquisition scan (MUGA) performed within 28 days of screening.
* Subject has laboratory abnormalities, or clinical evidence of disseminated intravascular coagulation, or ongoing history of coagulation disorder manifested by bleeding or clotting.
* Subject has an active uncontrolled infection.
* Subject is known to have human immunodeficiency virus infection.
* Subject has active hepatitis B or C or other active hepatic disorder.
* Subject has any condition which makes the subject unsuitable for study participation.
* Subject has a known or suspected hypersensitivity to bovine-derived protein or has suspected hypersensitivity to any ingredients of ASP7517.
* Subject is eligible for HSCT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (16):
- United States (3):
  - City of Hope, Duarte, California
  - Memorial Healthcare System-West, Pembroke Pines, Florida
  - NYU Langone Health, New York, New York
- Japan (13):
  - Site JP81005, Nagoya, Aichi-ken
  - Site JP81016, Matsuyama, Ehime
  - Site JP81009, Yoshida-gun, Fukui
  - Site JP81004, Maebashi, Gunma
  - Site JP81007, Kobe, Hyōgo
  - Site JP81013, Isehara, Kanagawa
  - Site JP81017, Sendai, Miyagi
  - Site JP81001, Shinagawa, Tokyo
  - Site JP81002, Fukuoka
  - Site JP81010, Gifu
  - Site JP81008, Okayama
  - Site JP81011, Osaka
  - Site JP81012, Osaka

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to plain language summary of the study on the Trial Results Summaries website. — https://ast.trialsummaries.com/Study/StudyDetails?id=14575&tenant=MT_AST_9011
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website. — https://www.clinicaltrials.astellas.com/study/7517-CL-0101/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with relapsed/refractory acute myeloid leukemia and relapsed/refractory higher risk myelodysplastic syndrome were enrolled in the study.
Pre-assignment Details: Participants who met all inclusion criteria and none of the exclusion criteria were enrolled in the study.
Period: Dose Escalation Phase (56 Days)
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Started | 6 | 5 | 8 | 0 | 0
Completed | 2 | 1 | 4 | 0 | 0
Not Completed | 4 | 4 | 4 | 0 | 0
Not completed — Progressive disease | 1 | 1 | 1 | 0 | 0
Not completed — Lack of Efficacy | 3 | 3 | 3 | 0 | 0
Period: Dose Expansion Phase (168 Days)
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Started | 0 | 0 | 0 | 12 | 12
Completed | 0 | 0 | 0 | 1 | 3
Not Completed | 0 | 0 | 0 | 11 | 9
Not completed — Miscellaneous | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 6 | 5
Not completed — Lack of Efficacy | 0 | 0 | 0 | 3 | 2
Not completed — Death | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) consisted of all participants who were enrolled and received at least one dose of study drug.
Groups:
- Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL: Participants with R/R AML and R/R higher risk MDS received IV infusion of ASP7517 (HEK293 transfected with encoding target WT-1) at a dose of 1x10^6 cells/mL at 4 to 6 mL/minute infusion rate on day 1 of each cycle for 2 doses (1 cycle= 28 days).
- Total: Total of all reporting groups
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL | Total
Number analyzed (Participants) | 6 | 5 | 8 | 12 | 12 | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.7 (3.8) | 76.2 (4.3) | 76.1 (2.5) | 72.8 (4.5) | 70.8 (7.7) | 73.0 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 4 | 4 | 15
  Male | 3 | 4 | 5 | 8 | 8 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 4 | 4 | 8 | 11 | 11 | 38
  Unknown or Not Reported | 2 | 1 | 0 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 5 | 8 | 10 | 9 | 38
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 2 | 3 | 5
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
ECOG Perfomance Status (PS) [Number; unit: Participants] — Number of participants with ECOG PS was reported and was measured on 6-point grade scale 0: Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory & able to carry out work of light or sedentary nature
  2. Ambulatory & capable of all self-care but unable to carry out any work activities. Up and about more than (>) 50% of waking hours
  3. Capable of only limited self-care, confined to bed or chair > 50% of waking hours
  4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair
  5. Dead
  Participants
    Grade 0 | 1 | 3 | 3 | 8 | 5 | 20
    Grade 1 | 5 | 2 | 4 | 2 | 6 | 19
    Grade 2 | 0 | 0 | 1 | 2 | 1 | 4
    Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
    Grade 4 | 0 | 0 | 0 | 0 | 0 | 0
    Grade 5 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT was defined as any of the following events that occurred within 28 days starting with the first dose on cycle 1 day 1 (C1D1) and that was considered to be related to study drug. DLT was defined as follows:
  * Grade 3 of more : non-hematologic AEs that are ≥ grade 3
  * Confirmed Hy's law case
  * New onset of grade 4 thrombocytopenia (with minimum of 2 grade worsening from baseline) within 24 hours of dosing
  * Prolonged myelosuppression, defined as absolute neutrophil count (ANC) < 500/microliter (μL) for more than 28 days off therapy and in the absence of evidence of active leukemia or MDS in the marrow or blood.
Time Frame: Day 1 up to 28 days
Population: The safety analysis set (SAF) consisted of all participants who were enrolled and received at least 1 dose of study drug.
  SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 4 | 4 | 6 | 9 | 11
participants | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) & Serious TEAE
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE could therefore be any unfavorable & unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An AE was considered "serious" if, it resulted in any of the following outcomes: results in death; is life-threatening; results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions; results in congenital anomaly, or birth defect; requires inpatient hospitalization; or leads to prolongation of hospitalization; other medically important events. TEAE was defined as an AE observed after starting administration of the study drug. TEAEs included both Serious and non-serious AEs.
Time Frame: From first dose up to 43 months
Population: SAF
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 6 | 5 | 8 | 12 | 12
participants
  TEAE | 5 | 5 | 6 | 12 | 10
  Serious TEAE | 1 | 4 | 2 | 8 | 5

3. Primary Outcome: Phase 2: Composite Complete Remission (CRc) Rate for Participants With R/R AML
Description: Percentage of participants with CRc was reported. CRc:defined as rate of all complete & incomplete remissions (CR + CR with incomplete platelet recovery [CRp] + CR with incomplete hematological recover [Cri]). CR: achieved morphologic leukemia-free state & their bone marrow was regenerating normal hematopoietic cells. If absolute neutrophil count (ANC) ≥ 1×10^9/L, platelet count (PC) ≥ 100×10^9/L, normal marrow differential < 5% blasts, & were red blood cell (RBC) and platelet transfusion independent (defined as 1 week without RBC transfusion & platelet transfusion prior to disease assessment). There was no evidence of extramedullary leukemia or Auer rods & blast counts in peripheral blood must be ≤ 2%. CRp: must achieve CR except for incomplete platelet recovery (< 100×10^9/L). CRi: must fulfil CR except for incomplete hematological recovery with residual neutropenia (ANC < 1×10^9/L), with or without complete platelet recovery. RBC and platelet transfusion independence not required.
Time Frame: From first dose up to 43 months
Population: FAS with available data was analyzed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Dose Escalation (Phase 1) (AML): ASP7517 1x10^6 Cells/mL: Participants with R/R AML received IV infusion of ASP7517 (HEK293 transfected with encoding target WT-1) at a dose of 1x10^6 cells/mL at 4 to 6 mL/minute infusion rate on day 1 of each cycle for 2 doses (1 cycle= 28 days).
- Dose Escalation (Phase 1) (AML): ASP7517 1x10^7 Cells/mL: Participants with R/R AML received IV infusion of ASP7517 (HEK293 transfected with encoding target WT-1) at a dose of 1x10^7 cells/mL at 4 to 6 mL/minute infusion rate on day 1 of each cycle for 2 doses (1 cycle= 28 days).
- Dose Escalation (Phase 1) (AML): ASP7517 1x10^8 Cells/mL: Participants with R/R AML received IV infusion of ASP7517 (HEK293 transfected with encoding target WT-1) at a dose of 1x10^8 cells/mL at 4 to 6 mL/minute infusion rate on day 1 of each cycle for 2 doses (1 cycle= 28 days).
Arm/Group | Dose Escalation (Phase 1) (AML): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1) (AML): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1) (AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 5 | 3 | 7 | 12
percentage of participants | 0.0 [0.0 to 45.1] | 0.0 [0.0 to 63.2] | 14.3 [0.7 to 52.1] | 8.3 [0.4 to 33.9]

4. Primary Outcome: Phase 2: Complete Remission + Bone Marrow Complete Remission + Partial Remission (CR + BM CR + PR) Rate for Participants With R/R Higher Risk MDS
Description: Percentage of participants with CR+BM CR+ PR was reported. CR, BM CR and PR achieved for minimum of 4 weeks; CR: bone marrow: ≤ 5% myeloblasts with normal maturation of all cell Lines, peripheral blood evaluation (hemoglobin (Hb) ≥ 11 g/dL, platelets ≥ 100 × 10^9/L, neutrophils ≥ 1.0 × 10^9/L, 0% blasts in blood)
  BM CR: bone marrow: ≤ 5% myeloblasts and decrease by ≥ 50% over pretreatment
  PR: achieved all CR criteria except bone marrow blasts decreased by ≥ 50% over pretreatment but still > 5%, cellularity and morphology not relevant.
Time Frame: From first dose up to 43 months
Population: FAS with available data was analyzed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Dose Escalation (Phase 1) (MDS): ASP7517 1x10^6 Cells/mL: Participants with R/R higher risk MDS received IV infusion of ASP7517 (HEK293 transfected with encoding target WT-1) at a dose of 1x10^6 cells/mL at 4 to 6 mL/minute infusion rate on day 1 of each cycle for 2 doses (1 cycle= 28 days).
- Dose Escalation (Phase 1) (MDS): ASP7517 1x10^7 Cells/mL: Participants with R/R higher risk MDS received IV infusion of ASP7517 (HEK293 transfected with encoding target WT-1) at a dose of 1x10^7 cells/mL at 4 to 6 mL/minute infusion rate on day 1 of each cycle for 2 doses (1 cycle= 28 days).
- Dose Escalation (Phase 1) (MDS): ASP7517 1x10^8 Cells/mL: Participants with R/R higher risk MDS received IV infusion of ASP7517 (HEK293 transfected with encoding target WT-1) at a dose of 1x10^8 cells/mL at 4 to 6 mL/minute infusion rate on day 1 of each cycle for 2 doses (1 cycle= 28 days).
Arm/Group | Dose Escalation (Phase 1) (MDS): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1) (MDS): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1) (MDS): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 1 | 2 | 1 | 12
percentage of participants | 100.0 [5.0 to 100.0] | 0.0 [0.0 to 77.6] | 0.0 [0.0 to 95.0] | 0.0 [0.0 to 22.1]

5. Primary Outcome: Number of Participants With ECOG Performance Status at Cycle 1(C1) Day2(D2)
Description: Number of participants with ECOG PS was reported. ECOG performance status was measured on a 6 point grade scale.
  0: Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  5. Dead.
Time Frame: C1D2
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 6 | 5 | 8 | 12 | 11
participants
  Grade 0 | 1 | 3 | 3 | 8 | 6
  Grade 1 | 5 | 2 | 4 | 2 | 4
  Grade 2 | 0 | 0 | 1 | 2 | 1
  Grade 3 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With ECOG Performance Status at C1D4
Description: as for outcome 5
Time Frame: C1D4
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 6 | 5 | 8 | 0 | 0
participants
  Grade 0 | 1 | 3 | 2 |  |
  Grade 1 | 5 | 2 | 5 |  |
  Grade 2 | 0 | 0 | 1 |  |
  Grade 3 | 0 | 0 | 0 |  |
  Grade 4 | 0 | 0 | 0 |  |
  Grade 5 | 0 | 0 | 0 |  |

7. Primary Outcome: Number of Participants With ECOG Performance Status at C1D8
Description: as for outcome 5
Time Frame: C1D8
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 6 | 5 | 8 | 12 | 12
participants
  Grade 0 | 1 | 3 | 2 | 8 | 4
  Grade 1 | 5 | 2 | 5 | 2 | 7
  Grade 2 | 0 | 0 | 1 | 2 | 1
  Grade 3 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With ECOG Performance Status at C1D11
Description: as for outcome 5
Time Frame: C1D11
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 5 | 8 | 0 | 0
participants
  Grade 0 |  | 3 | 2 |  |
  Grade 1 |  | 2 | 5 |  |
  Grade 2 |  | 0 | 1 |  |
  Grade 3 |  | 0 | 0 |  |
  Grade 4 |  | 0 | 0 |  |
  Grade 5 |  | 0 | 0 |  |

9. Primary Outcome: Number of Participants With ECOG Performance Status at C1D15
Description: as for outcome 5
Time Frame: C1D15
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 5 | 5 | 8 | 12 | 12
participants
  Grade 0 | 2 | 3 | 3 | 5 | 5
  Grade 1 | 3 | 2 | 4 | 4 | 5
  Grade 2 | 0 | 0 | 1 | 2 | 2
  Grade 3 | 0 | 0 | 0 | 1 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With ECOG Performance Status at C1D18
Description: as for outcome 5
Time Frame: C1D18
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 5 | 7 | 0 | 0
participants
  Grade 0 |  | 3 | 3 |  |
  Grade 1 |  | 2 | 3 |  |
  Grade 2 |  | 0 | 1 |  |
  Grade 3 |  | 0 | 0 |  |
  Grade 4 |  | 0 | 0 |  |
  Grade 5 |  | 0 | 0 |  |

11. Primary Outcome: Number of Participants With ECOG Performance Status at C1D22
Description: as for outcome 5
Time Frame: C1D22
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 4 | 5 | 7 | 9 | 8
participants
  Grade 0 | 2 | 3 | 3 | 6 | 3
  Grade 1 | 2 | 2 | 3 | 1 | 4
  Grade 2 | 0 | 0 | 1 | 1 | 1
  Grade 3 | 0 | 0 | 0 | 1 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Participants With ECOG Performance Status at C1D25
Description: as for outcome 5
Time Frame: C1D25
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 4 | 7 | 0 | 0
participants
  Grade 0 |  | 2 | 3 |  |
  Grade 1 |  | 2 | 3 |  |
  Grade 2 |  | 0 | 1 |  |
  Grade 3 |  | 0 | 0 |  |
  Grade 4 |  | 0 | 0 |  |
  Grade 5 |  | 0 | 0 |  |

13. Primary Outcome: Number of Participants With ECOG Performance Status at C2D1
Description: as for outcome 5
Time Frame: C2D1
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 4 | 4 | 6 | 8 | 9
participants
  Grade 0 | 1 | 1 | 2 | 6 | 4
  Grade 1 | 3 | 3 | 3 | 0 | 5
  Grade 2 | 0 | 0 | 0 | 2 | 0
  Grade 3 | 0 | 0 | 1 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0

14. Primary Outcome: Number of Participants With ECOG Performance Status at C2D2
Description: as for outcome 5
Time Frame: C2D2
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 4 | 3 | 6 | 8 | 8
participants
  Grade 0 | 1 | 1 | 3 | 5 | 4
  Grade 1 | 3 | 2 | 2 | 0 | 4
  Grade 2 | 0 | 0 | 0 | 3 | 0
  Grade 3 | 0 | 0 | 1 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0

15. Primary Outcome: Number of Participants With ECOG Performance Status at C2D4
Description: as for outcome 5
Time Frame: C2D4
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 4 | 2 | 6 | 0 | 0
participants
  Grade 0 | 1 | 0 | 3 |  |
  Grade 1 | 3 | 2 | 2 |  |
  Grade 2 | 0 | 0 | 0 |  |
  Grade 3 | 0 | 0 | 1 |  |
  Grade 4 | 0 | 0 | 0 |  |
  Grade 5 | 0 | 0 | 0 |  |

16. Primary Outcome: Number of Participants With ECOG Performance Status at C2D8
Description: as for outcome 5
Time Frame: C2D8
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 4 | 2 | 6 | 8 | 6
participants
  Grade 0 | 2 | 0 | 2 | 6 | 3
  Grade 1 | 2 | 2 | 3 | 1 | 3
  Grade 2 | 0 | 0 | 1 | 1 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0

17. Primary Outcome: Number of Participants With ECOG Performance Status at C2D15
Description: as for outcome 5
Time Frame: C2D15
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 3 | 1 | 5 | 6 | 7
participants
  Grade 0 | 2 | 0 | 2 | 5 | 3
  Grade 1 | 1 | 1 | 2 | 1 | 4
  Grade 2 | 0 | 0 | 1 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0

18. Primary Outcome: Number of Participants With ECOG Performance Status at C2D22
Description: as for outcome 5
Time Frame: C2D22
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 3 | 1 | 5 | 5 | 7
participants
  Grade 0 | 2 | 0 | 3 | 3 | 3
  Grade 1 | 1 | 1 | 1 | 1 | 4
  Grade 2 | 0 | 0 | 1 | 1 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0

19. Primary Outcome: Number of Participants With ECOG Performance Status at C3D1
Description: as for outcome 5
Time Frame: C3D1
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 0 | 0 | 3 | 7
participants
  Grade 0 |  |  |  | 2 | 3
  Grade 1 |  |  |  | 0 | 4
  Grade 2 |  |  |  | 1 | 0
  Grade 3 |  |  |  | 0 | 0
  Grade 4 |  |  |  | 0 | 0
  Grade 5 |  |  |  | 0 | 0

20. Primary Outcome: Number of Participants With ECOG Performance Status at C3D15
Description: as for outcome 5
Time Frame: C3D15
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 0 | 0 | 3 | 6
participants
  Grade 0 |  |  |  | 1 | 3
  Grade 1 |  |  |  | 2 | 3
  Grade 2 |  |  |  | 0 | 0
  Grade 3 |  |  |  | 0 | 0
  Grade 4 |  |  |  | 0 | 0
  Grade 5 |  |  |  | 0 | 0

21. Primary Outcome: Number of Participants With ECOG Performance Status at C4D1
Description: as for outcome 5
Time Frame: C4D1
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 0 | 0 | 3 | 5
participants
  Grade 0 |  |  |  | 1 | 2
  Grade 1 |  |  |  | 2 | 3
  Grade 2 |  |  |  | 0 | 0
  Grade 3 |  |  |  | 0 | 0
  Grade 4 |  |  |  | 0 | 0
  Grade 5 |  |  |  | 0 | 0

22. Primary Outcome: Number of Participants With ECOG Performance Status at C4D15
Description: as for outcome 5
Time Frame: C4D15
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 0 | 0 | 2 | 4
participants
  Grade 0 |  |  |  | 1 | 2
  Grade 1 |  |  |  | 1 | 2
  Grade 2 |  |  |  | 0 | 0
  Grade 3 |  |  |  | 0 | 0
  Grade 4 |  |  |  | 0 | 0
  Grade 5 |  |  |  | 0 | 0

23. Primary Outcome: Number of Participants With ECOG Performance Status at C5D1
Description: as for outcome 5
Time Frame: C5D1
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 0 | 0 | 2 | 5
participants
  Grade 0 |  |  |  | 1 | 2
  Grade 1 |  |  |  | 1 | 3
  Grade 2 |  |  |  | 0 | 0
  Grade 3 |  |  |  | 0 | 0
  Grade 4 |  |  |  | 0 | 0
  Grade 5 |  |  |  | 0 | 0

24. Primary Outcome: Number of Participants With ECOG Performance Status at C5D15
Description: as for outcome 5
Time Frame: C5D15
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 5
participants
  Gade 0 |  |  |  | 1 | 2
  Grade 1 |  |  |  | 0 | 3
  Grade 2 |  |  |  | 0 | 0
  Grade 3 |  |  |  | 0 | 0
  Grade 4 |  |  |  | 0 | 0
  Grade 5 |  |  |  | 0 | 0

25. Primary Outcome: Number of Participants With ECOG Performance Status at C6D1
Description: as for outcome 5
Time Frame: C6D1
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 3
participants
  Grade 0 |  |  |  | 0 | 0
  Grade 1 |  |  |  | 1 | 3
  Grade 2 |  |  |  | 0 | 0
  Grade 3 |  |  |  | 0 | 0
  Grade 4 |  |  |  | 0 | 0
  Grade 5 |  |  |  | 0 | 0

26. Primary Outcome: Number of Participants With ECOG Performance Status at C6D15
Description: as for outcome 5
Time Frame: C6D15
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 2
participants
  Grade 0 |  |  |  | 0 | 1
  Grade 1 |  |  |  | 1 | 1
  Grade 2 |  |  |  | 0 | 0
  Grade 3 |  |  |  | 0 | 0
  Grade 4 |  |  |  | 0 | 0
  Grade 5 |  |  |  | 0 | 0

27. Primary Outcome: Number of Participants With ECOG Performance Status at End of Treatment (EOT) (Dose Escalation Phase)
Description: Number of participants with ECOG PS was reported. ECOG performance status was measured on a 6 point grade scale.
  0: Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  5. Dead.
  EOT was calculated as last dose plus 7 days.
Time Frame: EOT (up to 63 Days)
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 5 | 3 | 8
participants
  Grade 0 | 3 | 1 | 3
  Grade 1 | 2 | 2 | 3
  Grade 2 | 0 | 0 | 1
  Grade 3 | 0 | 0 | 1
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

28. Primary Outcome: Number of Participants With ECOG Performance Status at EOT (Dose Expansion Phase)
Description: as for outcome 27
Time Frame: EOT (up to 175 days)
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 11 | 10
participants
  Grade 0 | 5 | 2
  Grade 1 | 1 | 6
  Grade 2 | 2 | 1
  Grade 3 | 1 | 1
  Grade 4 | 2 | 0
  Grade 5 | 0 | 0

29. Primary Outcome: Number of Participants With ECOG Performance Status at Observation Period (OP) (Week 2)
Description: Number of participants with ECOG PS was reported. ECOG performance status was measured on a 6 point grade scale.
  0: Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  5. Dead.
  OP was the period observed after the last dose.
Time Frame: OP (week 2)
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 1 | 0 | 0 | 2
participants
  Grade 0 |  | 0 |  |  | 0
  Grade 1 |  | 1 |  |  | 2
  Grade 2 |  | 0 |  |  | 0
  Grade 3 |  | 0 |  |  | 0
  Grade 4 |  | 0 |  |  | 0
  Grade 5 |  | 0 |  |  | 0

30. Primary Outcome: Number of Participants With ECOG Performance Status at OP (Week 4)
Description: as for outcome 29
Time Frame: OP (week 4)
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 2
participants
  Grade 0 | 1 |  |  |  | 0
  Grade 1 | 0 |  |  |  | 2
  Grade 2 | 0 |  |  |  | 0
  Grade 3 | 0 |  |  |  | 0
  Grade 4 | 0 |  |  |  | 0
  Grade 5 | 0 |  |  |  | 0

31. Primary Outcome: Number of Participants With ECOG Performance Status at OP (Week 6)
Description: as for outcome 29
Time Frame: OP (week 6)
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2
participants
  Grade 0 |  |  |  |  | 0
  Grade 1 |  |  |  |  | 2
  Grade 2 |  |  |  |  | 0
  Grade 3 |  |  |  |  | 0
  Grade 4 |  |  |  |  | 0
  Grade 5 |  |  |  |  | 0

32. Primary Outcome: Number of Participants With ECOG Performance Status at OP (Week 8)
Description: as for outcome 29
Time Frame: OP (week 8)
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 2
participants
  Grade 0 | 1 |  |  |  | 0
  Grade 1 | 0 |  |  |  | 2
  Grade 2 | 0 |  |  |  | 0
  Grade 3 | 0 |  |  |  | 0
  Grade 4 | 0 |  |  |  | 0
  Grade 5 | 0 |  |  |  | 0

33. Primary Outcome: Number of Participants With ECOG Performance Status at OP (Week 10)
Description: as for outcome 29
Time Frame: OP (week 10)
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2
participants
  Grade 0 |  |  |  |  | 0
  Grade 1 |  |  |  |  | 2
  Grade 2 |  |  |  |  | 0
  Grade 3 |  |  |  |  | 0
  Grade 4 |  |  |  |  | 0
  Grade 5 |  |  |  |  | 0

34. Primary Outcome: Number of Participants With ECOG Performance Status at OP (Week 12)
Description: as for outcome 29
Time Frame: OP (week 12)
Population: SAF with available data was analyzed
Measure: Number; unit: participants
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
participants
  Grade 0 |  |  |  |  | 0
  Grade 1 |  |  |  |  | 1
  Grade 2 |  |  |  |  | 0
  Grade 3 |  |  |  |  | 0
  Grade 4 |  |  |  |  | 0
  Grade 5 |  |  |  |  | 0

35. Secondary Outcome: Duration of Remission (DR) for Participants With R/R AML
Description: DR for AML: included duration of CRc, duration of CR/complete remission with partial hematologic recovery (CRh), duration of CRh, duration of CR, and duration of response (i.e., CRc + PR).
  CRh: achieved marrow blasts < 5%, partial hematologic recovery ANC ≥ 0.5 × 10^9/L and platelets ≥ 50 × 10^9/L, no evidence of extramedullary leukemia and cannot be classified as CR. The blast counts in peripheral blood was ≤ 2%.
  PR for AML; achieved bone marrow regenerating normal hematopoietic cells with evidence of peripheral recovery with no (or only a few regenerating) circulating blasts with decrease of at least 50% in the percentage of blasts in bone marrow aspirate with total marrow blasts between 5% and 25%. Value ≤ 5% blasts was considered PR if Auer rods were present. No evidence of extramedullary leukemia.
  CR, CRc were defined in outcome measure #3. Kaplan Meier (KM) Estimate was used.
Time Frame: From first response up to 43 months
Population: Response Analysis Set (RAS) included FAS participants and had at least 1 post baseline primary efficacy measurement. As per change in the planned analysis, the dose level utilized during the expansion phase was the RP2D, which was carefully selected from the dose escalation phase and a pooled population was used to estimate time-to-event efficacy endpoints for a comprehensive overview of the treatment's effectiveness.
Measure: Median (90% Confidence Interval); unit: days
Groups:
- Dose Escalation and Expansion Phase (AML): ASP7517 1x10^8 Cells/mL: Participants with R/R AML received IV infusion of ASP7517 (HEK293 transfected with encoding target WT-1) at a dose of 1x10^8 cells/mL at 4 to 6 mL/minute infusion rate on day 1 of each cycle (escalation phase: 2 doses and expansion phase: 6 doses) (1 cycle= 28 days).
Arm/Group | Dose Escalation (Phase 1) (AML): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1) (AML): ASP7517 1x10^7 Cells/mL | Dose Escalation and Expansion Phase (AML): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 3 | 3 | 15
days
  Duration of CRc: number analyzed (Participants) | 0 | 0 | 2
  Duration of CRc |  |  | 15.0 [15.0 to 15.0]
  Duration of CR/CRh: number analyzed (Participants) | 0 | 0 | 0
  Duration of CRh: number analyzed (Participants) | 0 | 0 | 0
  Duration of CR: number analyzed (Participants) | 0 | 0 | 0
  Duration of response: number analyzed (Participants) | 0 | 0 | 5
  Duration of response |  |  | 55.0 [15.0 to 55.0]

36. Secondary Outcome: Duration of Remission (DR) for Participants With R/R Higher Risk MDS
Description: DR for MDS: included duration of CR and duration of response (i.e., CR + BM CR + PR).
  CR, BM CR and PR achieved for minimum of 4 weeks; CR: bone marrow: ≤ 5% myeloblasts with normal maturation of all cell Lines, peripheral blood evaluation (hemoglobin (Hb) ≥ 11 g/dL, platelets ≥ 100 × 10^9/L, neutrophils ≥ 1.0 × 10^9/L, 0% blasts in blood)
  BM CR: bone marrow: ≤ 5% myeloblasts and decrease by ≥ 50% over pretreatment
  PR: achieved all CR criteria except bone marrow blasts decreased by ≥ 50% over pretreatment but still > 5%, cellularity and morphology not relevant. KM Estimate was used.
Time Frame: From first response up to 43 months
Population: RAS As per change in the planned analysis, the dose level utilized during the expansion phase was the RP2D, which was carefully selected from the dose escalation phase and a pooled population was used to estimate time-to-event efficacy endpoints for a comprehensive overview of the treatment's effectiveness.
Measure: Median (90% Confidence Interval); unit: days
Groups:
- Dose Escalation and Expansion Phase (MDS): ASP7517 1x10^8 Cells/mL: Participants with R/R higher risk MDS received IV infusion of ASP7517 (HEK293 transfected with encoding target WT-1) at a dose of 1x10^8 cells/mL at 4 to 6 mL/minute infusion rate on day 1 of each cycle (escalation phase: 2 doses and expansion phase: 6 doses) (1 cycle= 28 days).
Arm/Group | Dose Escalation (Phase 1) (MDS): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1) (MDS): ASP7517 1x10^7 Cells/mL | Dose Escalation and Expansion Phase (MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 1 | 1 | 11
days
  Duration of Response: number analyzed (Participants) | 1 | 0 | 0
  Duration of Response | 2.0 [NA to NA] — Data was not estimable as only 1 participant was evaluable. |  |
  Duration of CR: number analyzed (Participants) | 0 | 0 | 0

37. Secondary Outcome: Event Free Survival (EFS)
Description: EFS was defined as the time from the date of first dose until the date of documented relapse, treatment failure or death from any cause within 30 days after the last dose of study drug (whichever occurred first earliest of [relapse date, treatment failure date, death date] - first dose date + 1). Relapse was defined as a reappearance of leukemic blasts in the peripheral blood (> 2%) or ≥ 5% blasts in the bone marrow aspirate not attributable to any other cause or reappearance or new appearance of extramedullary leukemia or reappearance of significant numbers of peripheral blasts and an increase in the percentage of blasts in the bone marrow aspirate to > 25% not attributable to any other cause or reappearance or new appearance of extramedullary leukemia. KM Estimate was used.
Time Frame: From first dose up to 43 months
Population: FAS As per change in the planned analysis, the dose level utilized during the expansion phase was the RP2D, which was carefully selected from the dose escalation phase and a pooled population was used to estimate time-to-event efficacy endpoints for a comprehensive overview of the treatment's effectiveness.
Measure: Median (90% Confidence Interval); unit: days
Groups:
- Dose Escalation (Phase 1) (MDS): ASP7517 1x10^6 Cells/m: Participants with R/R higher risk MDS received IV infusion of ASP7517 (HEK293 transfected with encoding target WT-1) at a dose of 1x10^6 cells/mL at 4 to 6 mL/minute infusion rate on day 1 of each cycle for 2 doses (1 cycle= 28 days).
- Dose Escalation and Expansion (MDS): ASP7517 1x10^8 Cells/mL: Participants with R/R higher risk MDS received IV infusion of ASP7517 (HEK293 transfected with encoding target WT-1) at a dose of 1x10^8 cells/mL at 4 to 6 mL/minute infusion rate on day 1 of each cycle (escalation phase: 2 doses and expansion phase: 6 doses) (1 cycle= 28 days).
Arm/Group | Dose Escalation (Phase 1) (AML): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1) (AML): ASP7517 1x10^7 Cells/mL | Dose Escalation and Expansion Phase (AML): ASP7517 1x10^8 Cells/mL | Dose Escalation (Phase 1) (MDS): ASP7517 1x10^6 Cells/m | Dose Escalation (Phase 1) (MDS): ASP7517 1x10^7 Cells/mL | Dose Escalation and Expansion (MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 5 | 3 | 19 | 1 | 2 | 13
days | 44.0 [12.0 to 81.0] | 32.0 [30.0 to 50.0] | 58.0 [38.0 to 71.0] | 30.0 [NA to NA] — Data was not estimable as only 1 participant was evaluable. | NA [23.0 to NA] — Data was not estimable less than 50% participant had events. | 63.0 [28 to 120]

38. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first dose until the date of death from any cause (death date - first dose date + 1). For a Participant who was not known to have died by the end of study follow-up, OS was censored at the date of last contact (date of last contact - first dose date + 1). KM Estimate was used.
Time Frame: From first dose up to 43 months
Population: as for outcome 37
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Dose Escalation (Phase 1) (AML): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1) (AML): ASP7517 1x10^7 Cells/mL | Dose Escalation and Expansion Phase (AML): ASP7517 1x10^8 Cells/mL | Dose Escalation (Phase 1) (MDS): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1) (MDS): ASP7517 1x10^7 Cells/mL | Dose Escalation and Expansion Phase (MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 5 | 3 | 19 | 1 | 2 | 13
days | 159.0 [110.0 to 482.0] | 343.0 [289.0 to 532.0] | 162.0 [83.0 to 316.0] | 883.0 [NA to NA] — Data was not estimable as only 1 participant was evaluable. | 88.5 [47.0 to 130.0] | 180.0 [82.0 to NA] — Data was not estimable less than 50% participant had events.

39. Secondary Outcome: CR for Participants With R/R AML
Description: Percentage of participants with CR was reported. CR: achieved morphologic leukemia-free state & their bone marrow was regenerating normal hematopoietic cells. If absolute neutrophil count (ANC) ≥ 1 × 10^9/L, platelet count (PC) ≥ 100 × 10^9/L, normal marrow differential < 5% blasts, & were red blood cell (RBC) and platelet transfusion independent (defined as 1 week without RBC transfusion & platelet transfusion prior to disease assessment). There was no evidence of extramedullary leukemia or Auer rods and blast counts in peripheral blood must be ≤ 2%.
Time Frame: From first dose up to 43 months
Population: FAS with available data was analyzed.
Measure: Number; unit: percentage of participants
Groups:
- Dose Expansion (Phase 2) (AML): ASP7517 1x10^8 Cells/mL: Participants with R/R AML received IV infusion of ASP7517 (HEK293 transfected with encoding target WT-1) at a dose of 1x10^8 cells/mL at 4 to 6 mL/minute infusion rate on day 1 of each cycle for 6 doses (1 cycle= 28 days).
Arm/Group | Dose Escalation (Phase 1) (AML): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1) (AML): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1) (AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2) (AML): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 5 | 3 | 7 | 12
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0

40. Secondary Outcome: Best Response (CRc + PR) Rates for Participants With R/R AML
Description: Percentage of participants with best response (CRc + PR) was reported. CRc was defined as rate of all complete and incomplete remissions (CR + CR with incomplete platelet recovery [CRp] + CR with incomplete hematological recover [Cri]). CR, CRp and CRi were defined in Outcome measure # 3.
  PR: achieved bone marrow regenerating normal hematopoietic cells with evidence of peripheral recovery with no (or only a few regenerating) circulating blasts with decrease of at least 50% in the percentage of blasts in bone marrow aspirate with total marrow blasts between 5% and 25%. Value ≤ 5% blasts was considered PR if Auer rods were present. No evidence of extramedullary leukemia.
Time Frame: From first dose up to 43 months
Population: FAS with available data was analyzed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation (Phase 1) (AML): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1) (AML): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1) (AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2) (AML): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 5 | 3 | 7 | 12
percentage of participants | 0.0 [0.0 to 45.1] | 0.0 [0.0 to 63.2] | 28.6 [5.3 to 65.9] | 25.0 [7.2 to 52.7]

41. Secondary Outcome: CRh for Participants With R/R AML
Description: Percentage of participants with CRh was reported. CRh: achieved marrow blasts < 5%, partial hematologic recovery ANC ≥ 0.5 × 10^9/L and platelets ≥ 50 × 10^9/L, no evidence of extramedullary leukemia and cannot be classified as CR. The blast counts in peripheral blood was ≤ 2%.
Time Frame: From first dose up to 43 months
Population: FAS with available data was analyzed
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation (Phase 1) (AML): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1) (AML): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1) (AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2) (AML): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 5 | 3 | 7 | 12
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0

42. Secondary Outcome: CR for Participants With R/R Higher Risk MDS
Description: Percentage of participants with CR was reported. CR: bone marrow: ≤ 5% myeloblasts with normal maturation of all cell Lines, peripheral blood evaluation (hemoglobin (Hb) ≥ 11 g/dL, platelets ≥ 100 × 10^9/L, neutrophils ≥ 1.0 × 10^9/L, 0% blasts in blood).
Time Frame: From first dose up to 43 months
Population: FAS with available data was analyzed.
Measure: Number; unit: percentage of participants
Groups:
- Dose Escalation (Phase 1) (MDS): ASP7517 1x10^7 Cells/mL: Participant with R/R higher risk MDS received IV infusion of ASP7517 (HEK293 transfected with encoding target WT-1) at a dose of 1x10^7 cells/mL at 4 to 6 mL/minute infusion rate on day 1 of each cycle for 2 doses (1 cycle= 28 days).
- Dose Expansion (Phase 2) (MDS): ASP7517 1x10^8 Cells/mL: Participants with R/R higher risk MDS received IV infusion of ASP7517 (HEK293 transfected with encoding target WT-1) at a dose of 1x10^8 cells/mL at 4 to 6 mL/minute infusion rate on day 1 of each cycle for 6 doses (1 cycle= 28 days).
Arm/Group | Dose Escalation (Phase 1) (MDS): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1) (MDS): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1) (MDS): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2) (MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 1 | 2 | 1 | 12
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0

43. Secondary Outcome: Hematologic Improvement (HI) for Participants With R/R Higher Risk MDS
Description: Percentage of participants with HI was reported. HI: One measurement of the following for at least 8 weeks without cytotoxic therapy:
  * HI-erythroid: Hb increase of ≥ 1.5 g/dL or RBC transfusions performed for Hb ≤ 9.0 g/dL)
  * HI-platelets (pre-treatment PC: >20 ×10^9/L platelet, absolute increase of ≥ 30 ×10^9/L and < 20 ×10^9/L, platelet absolute increase of > 20 ×10^9/L and ≥ 100% increase from pre-treatment level
  * HI-neutrophils (increase of ≥ 100% from pre-treatment level and an absolute increase of > 0.5 ×10^9/L)
Time Frame: From first dose up to 43 months
Population: FAS with available data was analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation (Phase 1) (MDS): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1) (MDS): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1) (MDS): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2) (MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 1 | 2 | 1 | 12
percentage of participants
  HI - Erythroid | 0.0 | 0.0 | 0.0 | 8.3
  HI - Platelets | 0.0 | 0.0 | 0.0 | 0.0
  HI - Neutrophils | 0.0 | 0.0 | 0.0 | 8.3

44. Secondary Outcome: Objective Response (OR) (CR + BM CR + PR + HI) Rates (ORR) for Participants With R/R Higher Risk MDS
Description: Percentage of participants with OR (CR + BM CR + PR + HI) was reported. CR, BM CR & PR achieved for minimum of 4 weeks.
  CR: BM: ≤ 5% myeloblasts with normal maturation of all cell Lines peripheral blood evaluation (Hb) ≥ 11 g/dL platelets ≥ 100 × 10^9/L, neutrophils ≥ 1.0 × 10^9/L, 0% blasts in blood) BM CR: bone marrow ≤ 5% myeloblasts & decrease by ≥ 50% over pretreatment. PR: achieved all CR criteria except bone marrow blasts decreased ≥ 50% over pretreatment but still > 5% cellularity and morphology not relevant.
  HI: One measurement of following for at least 8 weeks without cytotoxic therapy.
  * HI-erythroid: Hb increase of ≥ 1.5 g/dL or RBC transfusions performed for Hb ≤ 9.0 g/dL)
  * HI-platelets (pre-treatment PC: >20 ×10^9/L platelet, absolute increase of ≥ 30 ×10^9/L and < 20 ×10^9/L, platelet absolute increase of > 20 ×10^9/L and ≥ 100% increase from pre-treatment level
  * HI-neutrophils (increase of ≥ 100% from pre-treatment level and an absolute increase of > 0.5 ×10^9/L)
Time Frame: From first dose up to 43 months
Population: FAS with available data was analyzed.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation (Phase 1) (MDS): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1) (MDS): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1) (MDS): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2) (MDS): ASP7517 1x10^8 Cells/mL
Number analyzed (Participants) | 1 | 2 | 1 | 12
percentage of participants | 100.0 [5.0 to 100.0] | 0.0 [0.0 to 77.6] | 0.0 [0.0 to 95.0] | 8.3 [0.4 to 33.9]

ADVERSE EVENTS:
Time Frame: From first dose up to 43 months
Description: SAF
Arm/Group | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL
All-Cause Mortality (participants affected / at risk) | 6/6 | 5/5 | 7/8 | 9/12 | 5/12
Serious Adverse Events (participants affected / at risk) | 1/6 | 4/5 | 2/8 | 8/12 | 5/12
Other Adverse Events (participants affected / at risk) | 5/6 | 4/5 | 6/8 | 10/12 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL (N=6) | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL (N=5) | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL (N=8) | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL (N=12) | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL (N=12)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | 3 (8) | 1 (1) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Device physical property issue (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation (Phase 1): ASP7517 1x10^6 Cells/mL (N=6) | Dose Escalation (Phase 1): ASP7517 1x10^7 Cells/mL (N=5) | Dose Escalation (Phase 1): ASP7517 1x10^8 Cells/mL (N=8) | Dose Expansion (Phase 2: AML): ASP7517 1x10^8 Cells/mL (N=12) | Dose Expansion (Phase 2: MDS): ASP7517 1x10^8 Cells/mL (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 2 (4)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 1 (2)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibrin D dimer increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (8)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Occipital neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement

DOCUMENTS (2):
  • Study Protocol (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/96/NCT04079296/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/96/NCT04079296/SAP_001.pdf